CLINICAL TRIAL: NCT03089840
Title: Assessing the Safety and Efficacy of a Portable Ex Vivo Oxygenated, Normothermic Liver Perfusion System (OrganOx Metra™ ) Prior to Liver Transplantation
Brief Title: Normothermic Liver Preservation Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00043239
Record Dates: First submitted 2017-03-11; First posted 2017-03-24 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: End Stage Liver Disease; Liver Diseases
Keywords: normothermic perfusion; liver transplantation
MeSH Terms: conditions — End Stage Liver Disease; Liver Diseases

STUDY DESIGN:
Intervention Model Description: Non-randomized, open-label, single arm, prospective trial using retrospective matched controls
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normothermic Machine Perfusion (OrganOx metra) (Experimental): Donor livers will be placed on the OrganOx metra device for normothermic perfusion before transplantation.
  Interventions: Device: OrganOx metra

INTERVENTIONS:
Device: OrganOx metra — Following the routine retrieval procedure at the donor hospital the liver will be flushed with cold preservation solution and prepared for cannulation. The donor organ is then placed on the OrganOx metra device and will be perfused with warmed solution. The OrganOx metra device containing the donor organ is then transported to the recipient transplant centre. The donor liver is then removed from the device and flushed with standard of care preservation solution. Alternatively, where more practical, the livers will be transported to the University of Alberta hospital with ≤ 6 hours of cold storage and then placed on the metra™ for ≥ 4 hours. Implantation and reperfusion of the liver proceed as per the usual practice of the recipient transplant centre.

SUMMARY:
This trial is to assess the safety and efficacy of normothermic machine perfusion (NMP) as an organ preservation method prior to transplantation using the OrganOx metra™ device.

DETAILED DESCRIPTION:
The standard approach for storage and transportation of livers for transplantation involves cold perfusion with Histidine-tryptophan-ketoglutarate (HTK) or alternative solutions, and storage in sterile bags surrounded by preservation solution in a box by ice. The prolonged cold ischemic injury substantially compounds pre-existing donor liver graft injury, further exacerbating potential risk for recipients. Normothermic perfusion may eliminate cold ischemic injury, and provide a unique opportunity to further assess ex vivo function of the most marginal organs before they are transplanted. Being able to select or eliminate organs in this manner would provide additional livers for transplantation while at the same time minimizing risk for recipients.

This non-randomized, open-label, single arm, prospective trial is to assess safety and preliminary efficacy of normothermic machine perfusion on livers accepted under standard and expanded criteria for standard liver transplantation (n=50). Following assessment of donor and recipient eligibility and confirmation of consent, the liver will be preserved on OrganOx metra™ either at the donor hospital or where more practical transported to the University of Alberta hospital with ≤ 6 hours of cold storage and then placed on the metra™ for ≥ 4 hours ('back to base' sub-analysis). At the end of preservation, the liver will be transplanted and the patient managed according to standard local practice and protocols. 100 anonymized patient data from the University of Alberta Hospital Liver Transplant database will be utilized for the matched controls. Enrolled subjects will participate in the study for 30 days (the accrued period to capture primary and secondary end-points: graft and patient survival, graft function, NMP perfusion parameters). Additional routine (non-research) biochemical and survival data will be collected and documented at 3, 6, 9 and 12 months post-transplant. Primary outcomes will be analyzed and reported 30 days following transplantation of the last subject in the study.

ELIGIBILITY:
Inclusion Criteria:

Recipient inclusion criteria:

Adult subjects (age ≥18 years); active on the waiting list for liver transplantation at the University of Alberta Hospital; informed/deferred consent provided.

Donor liver inclusion criteria:

Whole livers from deceased donors ≥ 40kg in weight, that are deemed suitable for transplantation as per local and international practice, and at the discretion of the transplanting surgeon.

Donor livers will be placed on the metra™ device either at the donor hospital, or where more practical, transported to the University of Alberta hospital with ≤ 6 hours of cold storage and then reperfused on metra™ for ≥ 4 hours ('back-to-base' sub-analysis).

Expanded criteria grafts may include, but not be restricted to the following graft qualities. Such grafts will only be transplanted at the recipient transplant surgeon's discretion, if judged to be safe and appropriate for that individual recipient.

Donation after Neurological Determination of Death (NDD) Expanded Criteria livers may include: ≥60% macro/micro steatosis; cold ischemia > 10 hours; combined steatosis 30-60% and >6hr cold storage; significant liver trauma.

Donation after Cardio-Circulatory Death (DCD) Expanded Criteria livers may include: Age up to 75; mild steatosis (30%); DCD offers from distant centres; warm time up to 60 min.

As per standard clinical practice, the on-call recipient transplant surgeon will evaluate donor and graft information, weigh the risks and benefits of graft utilization for a particular recipient, and make the final decision about whether or not to proceed to transplantation. Based on preliminary experience with the metraTM, perfusion parameters may additionally be considered in reaching a decision:

* Normal, stable portal vein flow (≥800-1000ml/minute) and artery flow (≥200ml/minute)
* Falling lactate levels
* Stable perfusate pH within the normal range (7.2 - 7.4) after bicarbonate correction
* Evenly perfused graft on the device

Exclusion Criteria:

Recipient exclusion criteria: Age less than 18 years, allergic to required components of the perfusion solution, refusal of informed consent.

Donor liver exclusion criteria: Livers from living donors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Graft survival rate | Day 30
  Graft survival rate

SECONDARY OUTCOMES:
Patient survival rate | Day 30
  Patient survival rate
Early Allograft Dysfunction (EAD) rate | Up to Day 7
  EAD rate
Peak aspartate transaminase (AST) levels | Up to Day 7
  Peak AST levels in the blood
Daily lactate levels | Up to Day 7
  Daily lactate levels in the blood
Perfusate AST levels | Day -1 and Day 0
  AST levels in perfusate blood
Perfusate alanine transaminase (ALT) levels | Day -1 and Day 0
  ALT levels in perfusate blood
Perfusate bilirubin levels | Day -1 and Day 0
  Bilirubin levels in perfusate blood
Perfusate lactate levels | Day -1 and Day 0
  Lactate levels in perfusate blood

CONTACTS AND LOCATIONS:
Overall Officials: James Shapiro, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada